CLINICAL TRIAL: NCT00373919
Title: The Effect of Erythromycin on Occurrence of Leaks From Cervical Esophageal-Gastric Anastomosis After Trans-Hiatal Esophagectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: erythro-esophagus
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2006-08

CONDITIONS: Esophagectomy; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

INTERVENTIONS:
Drug: intravenous (IV) administration of erythromycin

SUMMARY:
Cervical anastomotic leak is one of the most common complications after trans-hiatal esophagectomy.

Hypothesis: An early post operative administration of a pro-kinetic dosage of erythromycin will reduce leak occurrence.

Design: This is a prospective, randomized, double blind, placebo controlled study.

Number of patients: 30.

Inclusion Criteria:

* Patients after trans-hiatal esophagectomy

Exclusion Criteria:

* Allergy to erythromycin
* Use of phenothiazine
* QT prolongation
* Liver function test (LFT) abnormalities
* Myasthenia gravis
* Cardiomyopathy

ELIGIBILITY:
Inclusion Criteria:

* Patients after trans-hiatal esophagectomy

Exclusion Criteria:

* Allergy to erythromycin
* Use of phenothiazine
* QT prolongation
* Liver function test (LFT) abnormalities
* Myasthenia gravis
* Cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Koram Klein, MD, Principal Investigator — Kaplan Medical Center